CLINICAL TRIAL: NCT03087565
Title: Urinary and Sexual Functions After Subtotal Versus Total Abdominal Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 162
Record Dates: First submitted 2017-03-11; First posted 2017-03-22 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Sexual Function Disturbances; Urinary Function Disorders
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subtotal hystrectomy (Active Comparator): Careful examination under anesthesia. Catheterization by N. 18 Foley's catheter . A transverse lower abdominal incision (Pfannenstiel incision) . the corpus is amputated just below the level of the isthmus and then the endocervical canal is electrocoagulated using monopolar electrocautery. The cervical stump is closed using vicryl 0 sutures.
  Intraoperative antibiotics The abdomen is closed in layers; the wound is covered with a sterile dressing. All specimens were sent for pathological examination .
  Interventions: Procedure: subtotal hystrectomy
- Total hyterectomy (Active Comparator): examination under anesthesia. Catheterization by N. 18 Foley's catheter A transverse lower abdominal incision (Pfannenstiel incision) The urinary bladder is dissected off the lower uterine segment of the uterus and cervix by blunt or sharp dissection. Blunt dissection is done . Sharp dissection using Metzenbaum scissors is performed in patients with previous cesarean sections Revision of all pedicles to ensure hemostasis. Intraoperative antibiotics The abdomen is closed in layers; the wound is covered with a sterile dressing. All specimens were sent for pathological examination .
  Interventions: Procedure: Total hystrectomy

INTERVENTIONS:
Procedure: subtotal hystrectomy — A transverse lower abdominal incision (Pfannenstiel incision) The corpus is amputated just below the level of the isthmus and then the endocervical canal is electrocoagulated using monopolar electrocautery. The cervical stump is closed using vicryl 0 sutures.
  Revision of all pedicles to ensure hemostasis. Intraoperative antibiotics . The abdomen is closed in layers; the wound is covered with a sterile dressing.
  Arms: subtotal hystrectomy
Procedure: Total hystrectomy — A transverse lower abdominal incision (Pfannenstiel incision) The urinary bladder is dissected off the lower uterine segment of the uterus and cervix by blunt or sharp dissection. Revision of all pedicles to ensure hemostasis.
  The abdomen is closed in layers; the wound is covered with a sterile dressing.
  Arms: Total hyterectomy

SUMMARY:
All hysterectomies were performed intrafascially using the clamp-cut-ligate method as described by (Jones, 2003);

Careful examination under anesthesia.

Catheterization by N. 18 Foley's catheter and its balloon Filled with 10-ml saline.A transverse lower abdominal incision (Pfannenstiel incision) ranging from 8-12 cm through which the abdomen is opened in layers.

During subtotal hysterectomy procedure, the corpus is amputated just below the level of the isthmus and then the endocervical canal is electrocoagulated using monopolar electrocautery. The cervical stump is closed using vicryl 0 sutures.

During total hysterectomy procedure, the urinary bladder is dissected off the lower uterine segment of the uterus and cervix by blunt or sharp dissection. Blunt dissection is done using a finger pushed gently against the cervix rather than against the bladder. Sharp dissection using Metzenbaum scissors is performed in patients with previous cesarean sections, with upward traction on the bladder peritoneum and the uterine fundus stretched tightly out of the pelvis, the tips of the Metzenbaum scissors rest lightly on the fascia overlying the cervix with small bites to develop a tissue plane, dissecting the bladder from the anterior cervix.

Revision of all pedicles to ensure hemostasis.

Intraoperative antibiotics (1 gm of a 3rd generation cephalosporin + 0.5 gm metronidazole).

The abdomen is closed in layers; the wound is covered with a sterile dressing. All specimens were sent for pathological examination in the pathology Unit.

DETAILED DESCRIPTION:
All hysterectomies were performed intrafascially using the clamp-cut-ligate method as described by (Jones, 2003);

Careful examination under anesthesia.

Catheterization by N. 18 Foley's catheter and its balloon Filled with 10-ml saline.

A transverse lower abdominal incision (Pfannenstiel incision) ranging from 8-12 cm through which the abdomen is opened in layers.

During subtotal hysterectomy procedure, the corpus is amputated just below the level of the isthmus and then the endocervical canal is electrocoagulated using monopolar electrocautery. . The cervical stump is closed using vicryl 0 sutures.

During total hysterectomy procedure, the urinary bladder is dissected off the lower uterine segment of the uterus and cervix by blunt or sharp dissection. Blunt dissection is done using a finger pushed gently against the cervix rather than against the bladder. Sharp dissection using Metzenbaum scissors is performed in patients with previous cesarean sections, with upward traction on the bladder peritoneum and the uterine fundus stretched tightly out of the pelvis, the tips of the Metzenbaum scissors rest lightly on the fascia overlying the cervix with small bites to develop a tissue plane, dissecting the bladder from the anterior cervix.

Revision of all pedicles to ensure hemostasis.

Intraoperative antibiotics (1 gm of a 3rd generation cephalosporin + 0.5 gm metronidazole).

The abdomen is closed in layers; the wound is covered with a sterile dressing. All specimens were sent for pathological examination in the pathology Unit.

Post-operative care;

After ensuring complete recovery, the patient was transferred to the ward with close follow up of the vital signs every 15 minutes till stable, then every 2 hours for 24 hours, then every 8 hours till discharge.

Postoperative antibiotics (1 gm of a 3rd generation cephalosporin + 0.5 gm metronidazole) were given eight hourly for 24 hours then stopped (Hager, 2003).

Postoperative analgesics (Non-steroidal anti-inflammatory drugs) were given eight hourly for 24 hours then if needed

Intravenous fluids were given for the 1st 8 hours postoperative and then fluid diet was allowed with early ambulation and deep breathing (Horowitz and Basil, 2003).

The urinary catheter was removed 24 hours postoperatively.

Upon discharge, the patients were advised to resume work and sexual intercourse only after 4 weeks . An appointment was given to the patients to be seen 6 months after the operation.

Pre- and post-operative evaluation

The patients were interviewed and examined preoperatively and 6 months postoperative.

I. Urinary function was evaluated before surgery and 6 months afterward using;

A. Subjective questionnaire to detect urinary Symptoms including:

1. Diurnal frequency of micturition (voids >6 times a day).
2. Nocturia (waking at night more than one time to void).
3. Urge urinary incontinence. (urine leakage related to a feeling of urgency).
4. Stress urinary incontinence. (urine leakage related to physical activity, coughing or sneezing).
5. Dysuria (stinging/burning sensation).
6. Hesitancy (difficulty in initiating micturition).
7. Reduction of the stream (compared to previous performance).
8. Sensation of incomplete bladder emptying.
9. Haematuria.

B. Physical examination:

Stress test: With the bladder near full, the patient was asked to cough vigorously while watching for leakage of urine .

Evaluate levator ani muscle function by asking the patient to tighten her "vaginal muscles".

C. Objective urodynamic studies: urodynamic evaluation was done for all participants in the study. All urodynamic studies were performed using ANDROMEDA M00101-2 ELLIPSE.

The following tests were done:

1. Filling cystometry; the following parameters were evaluated and compared ;

   First desire to void (The point at which the woman first experiences an awareness of the need to empty her bladder).

   Maximum cystometric capacity (The point at which the woman can delay micturition no longer).

   Maximum detrusor pressure reached during filling phase.
2. Uroflowmetry:

Where the maximum flow rate and the residual volume were identified.

Method

1. The patient presented with a symptomatically full bladder. She voided spontaneously in a uroflow chair. Maximum flow rate and postvoid residual urine volume were obtained via a transurethral catheter.
2. The microtransducer catheters were connected to the appropriate cables and to the tubing from the water pump.
3. With the patient in the supine position on a urodynamic chair, the abdominal catheter was placed into the vagina . A dual microtransducer 6-French catheter with a filling port was then placed into the bladder . The patient was moved to a sitting position.
4. After the catheters were appropriately placed, the subtraction was checked by asking the patient to cough. Cough-induced pressure spikes should be seen on the Pves and Pabd channels, but not on the true detrusor pressure channel.
5. The urinary bladder was filled with normal saline at room temperature with a filling rate 50-100 ml/min. First desire to void and strong desire to void were recorded. Throughout the filling portion of the examination, the patient was asked to perform provocative activities, such as coughing and straining. The external urethral meatus was constantly observed for any involuntary urine loss.

Sexual function: The patients were interviewed before surgery and 6 months afterward and sexual function was evaluated using a subjective questionnaire measuring the following sexual variables :

1. Libido (desire): It is described as perceiving sexual desire once a week or more, which is a subjective feeling state.
2. Frequency of intercourse (once a week or more).
3. Dyspareunia (painful coitus).
4. Frequency of orgasm: the most intense pleasure followed by sudden release of the tension that has built up during excitement. It is described as (always or often).
5. Sense of vaginal dryness.
6. Satisfaction with sexual life (satisfied-not satisfied).

The patients were allowed to resume sexual intercourse 4 weeks after the operation.

Data collection included:

1. Postoperative recording of operation time, intra-operative blood transfusion (if needed), length of hospital stay, and pathology of the removed uterus.
2. Postoperative complications including pyrexia, vault haematoma, wound haematoma, wound infection, vaginal bleeding, need for blood transfusion, postoperative pain, cervical stump prolapse, and vaginal vault prolapse.

ELIGIBILITY:
Inclusion Criteria:

1. An age over 35 and below 50 years.
2. Menstruating women.
3. No symptomatic uterine prolapse. .
4. Normal cervical smears.
5. Benign lesions.
6. Active sexual life.
7. Functioning ovaries.

Exclusion Criteria:

1. Known endometriosis.
2. Overt neurological or psychiatric disorder.
3. Candidate for vaginal hysterectomy.
4. Use of hormone replacement therapy.
5. Oophorectomy.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Filling cystometry | 6 months after operation
  The patient presented with a symptomatically full bladder. She voided spontaneously in a uroflow chair. Maximum flow rate and postvoid residual urine volume were obtained via a transurethral catheter. The microtransducer catheters were connected to the appropriate cables and to the tubing from the water pump. With the patient in the supine position on a urodynamic chair, the abdominal catheter was placed into the vagina. A dual microtransducer 6-French catheter with a filling port was then placed into the bladder. The patient was moved to a sitting position. After the catheters were appropriately placed, the subtraction was checked by asking the patient to cough. Cough-induced pressure spikes should be seen on the Pves and Pabd channels, but not on the true detrusor pressure channel.
Uroflowmetry | 6 months after operation
  The urinary bladder was filled with normal saline at room temperature with a filling rate 50-100 ml/min. First desire to void and strong desire to void were recorded. Throughout the filling portion of the examination, the patient was asked to perform provocative activities, such as coughing and straining. The external urethral meatus was constantly observed for any involuntary urine loss.

SECONDARY OUTCOMES:
Sexual functions | 6 months after operation
  Satisfaction with sexual life (satisfied-not satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes